CLINICAL TRIAL: NCT05951556
Title: Individualizing Home Use of an Electroencephalographic or EEG-based Brain-computer Interface (BCI) Using Telemedicine
Brief Title: Telehealth Implementation of Brain-Computer Interface
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Albany Stratton VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Colin Franz, Attending MD, Principal investigator, Shirley Ryan AbilityLab
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ShirleyRyanAbilityLab
Record Dates: First submitted 2022-05-04; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Amyotrophic Lateral Sclerosis; Stroke
Keywords: locked in syndrome
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Stroke; Locked-In Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be provided with device; telehealth appts will be utilized to direct setup and usage of the device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- All Participants (Experimental): All Participants will receive trial device and will be trained (via Telehealth) in its use.
  Interventions: Device: Use of BCI

INTERVENTIONS:
Device: Use of BCI — Clients will utilize BCI with training to communicate wants and needs

SUMMARY:
Determine if Telehealth intervention can allow/empower a caregiver (who is untrained) to effectively implement and utilize a Brain-Computer Interface for communication with a participant who is "Locked in" following progression of Amyotrophic Lateral Sclerosis and other conditions.

DETAILED DESCRIPTION:
People with Amyotrophic Lateral Sclerosis (ALS) or other conditions such as a pontine stroke may develop a condition called Locked In Syndrome (LIS) where they are unable to use alternative communication strategies such as eyegaze to allow for communication for social needs or instruction to caregivers. Brain-Computer Interface (BCI) devices have been shown in the laboratory to allow participants to effectively communicate needs and engage in social communication. However, translation of this research to the home environment has been limited. In order to be a functional option for people to utilize, BCI needs to be much easier to set up and operate.

This study is designed to determine if telehealth intervention is sufficient to allow an untrained caregiver to set up and maintain a BCI for a person with a long-term communication difficulty given LIS.

Participants will receive a computer and associated hardware to allow for set up of the BCI. Videoconference support will be provided by the research team to allow the client and caregiver to set up the device in their home. Participants will hopefully be able to use the device to generate novel communication related to their care and engage in social needs with caregivers and/or family members. Communication that is generated will be logged and times that the participant is engaged in use of the BCI when not under direct support by the researchers will also be monitored.

The hypothesis is that telehealth support will be sufficient to allow for setting up the computer. If this is true, this will make it much easier for a client to engage in use of a BCI to allow for that communication versus the current need of traveling to a clinic or other specialized setting.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis leading to severe communication impairment

Exclusion Criteria:

-

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2024-07-05 (Estimated); Study Completion 2024-07-05 (Estimated)

PRIMARY OUTCOMES:
Log of communication | From date of enrollment in study until the date of discontinuation of the intervention, whichever came first, assessed up to 100 months
  Logs of any communication will be kept by monitoring number of accurate selections while utilizing the BCI.

CONTACTS AND LOCATIONS:
Overall Officials: Colin Franz, MD, Principal Investigator — SRALAB
Locations (1):
- ShirleyRyan AbilityLab, Chicago, Illinois, United States